CLINICAL TRIAL: NCT03565315
Title: VRC 610: Phase I Safety and Pharmacokinetics Study to Evaluate a Human Monoclonal Antibody (MAB) VRC-HIVMAB095-00-AB (10E8VLS) Administered Alone or Concurrently With MAB VRC-HIVMAB075-00-AB (VRC07-523LS) Via Subcutaneous Injection in Healthy Adults
Brief Title: Phase I Study to Evaluate a Human Monoclonal Antibody (MAb) 10E8VLS Administered Alone or Concurrently With MAb VRC07-523LS Via Subcutaneous Injection in Healthy Adults
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor/PI voluntarily paused and stopped study after observing several Grade 2 and Grade 3 redness local reactogenicity reactions at 10E8VLS injection sites
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 180113; 18-I-0113 (Other: NIH)
Record Dates: First submitted 2018-06-19; First posted 2018-06-21 (Actual); Results first posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Healthy Adult Immune Response
Keywords: HIV Prevention; Broadly Neutralizing Monoclonal Antibodies; First in Human Study; Anti-Drug Antibody Response to 10E8VLS or VRC07-523LS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: 10E8VLS (5 mg/kg) SC Single Dose Group (Experimental): 10E8VLS (5 mg/kg) administered by the subcutaneous (SC) route (Day 0)
  Interventions: Biological: VRC-HIVMAB095-00-AB (10E8VLS)
- Group 2: 10E8VLS (5 mg/kg) SC Multiple Dose Group* (*Only One Dose Received) (Experimental): 10E8VLS (5 mg/kg) administered by the SC route (Day 0, Week 12*, Week 24*)
  *Participants received only one product administration on Day 0 because of the voluntary study pause and termination by the IND Sponsor/PI decision.
  Interventions: Biological: VRC-HIVMAB095-00-AB (10E8VLS)
- Group 3: 10E8VLS+VRC07-523LS (5 mg/kg each) SC Single Dose Group (Experimental): 10E8VLS (5 mg/kg)+VRC07-523LS (5 mg/kg) administered by the SC route (Day 0)
  Interventions: Biological: VRC-HIVMAB095-00-AB (10E8VLS); Biological: VRC-HIVMAB075-00-AB (VRC07-523LS)
- Group 4: 10E8VLS+VRC07-523LS (5 mg/kg each) SC Multiple Dose Group* (*Only One Dose Received) (Experimental): 10E8VLS (5 mg/kg)+VRC07-523LS (5 mg/kg) administered by the SC route (Day 0, Week 12*, Week 24*)
  *Participants received only one product administration on Day 0 because of the voluntary study pause and termination by the IND Sponsor/PI decision.
  Interventions: Biological: VRC-HIVMAB095-00-AB (10E8VLS); Biological: VRC-HIVMAB075-00-AB (VRC07-523LS)

INTERVENTIONS:
Biological: VRC-HIVMAB095-00-AB (10E8VLS) — 10E8VLS is an investigational Monoclonal Antibody targeted to the membrane proximal external region and proximal viral membrane lipid region of HIV-1.
Biological: VRC-HIVMAB075-00-AB (VRC07-523LS) — VRC07-523LS is an investigational Monoclonal Antibody targeted to the CD4 binding site of HIV-1.
  Arms: Group 3: 10E8VLS+VRC07-523LS (5 mg/kg each) SC Single Dose Group; Group 4: 10E8VLS+VRC07-523LS (5 mg/kg each) SC Multiple Dose Group* (*Only One Dose Received)

SUMMARY:
Background:

Human immunodeficiency virus (HIV) infection is a serious disease. There is no cure or vaccine to prevent infection. Using antibodies might be a good way to treat or prevent HIV. Antibodies are naturally made by the body to fight germs. Researchers want to test if two antibodies made artificially in a lab can help to prevent HIV infection. The antibodies are 10E8VLS and VRC07-523LS.

Objective:

To see if 10E8VLS and VRC07-523LS are safe and well-tolerated and how long they stay in the blood.

Eligibility:

Healthy adults ages 18-60

Design:

Volunteers were screened in another protocol.

Participants were enrolled in 1 of 4 groups:

Group 1 participants were enrolled to receive 1 dose of 10E8VLS.

Group 2 participants were enrolled to receive 3 doses of 10E8VLS.

Group 3 participants were enrolled to receive 1 dose of both 10E8VLS and VRC07-523LS.

Group 4 participants were enrolled to receive 3 doses of both 10E8VLS and VRC07-523LS.

Participants in Groups 1 and 3 were expected to be enrolled about 13 visits over 24 weeks.

Participants in Groups 2 and 4 were expected to be enrolled about 26 visits over 48 weeks.

Participants were weighed before each dose. Women may have had a pregnancy test. Participants had blood collected.

A small needle injected each dose into fatty tissue of the belly, upper arm, or thigh. Participants received between 1 and 8 injections per dose depending on their weight. Heavier participants received more injections.

Participants received a ruler and thermometer. They checked their temperature for 3 days after injection(s) and measured any redness, swelling, or bruising at the injection site.

At non-injection visits, participants had blood drawn and were checked for health changes or problems.

DETAILED DESCRIPTION:
VRC 610:

A Phase I Safety and Pharmacokinetics Study to Evaluate a Human Monoclonal Antibody (MAB) VRC-HIVMAB095-00-AB (10E8VLS) Administered Alone or Concurrently with MAB VRC-HIVMAB075-00-AB (VRC07-523LS) Via Subcutaneous Injection in Healthy Adults

Study Design:

This first-in-human, open-label study evaluated MAb 10E8VLS (VRC-HIVMAB095-00-AB) administered alone or concurrently (i.e., at the same visit) with MAb VRC07-523LS (VRC-HIVMAB075-00-AB) in healthy adults ages 18 to 60. The primary hypothesis was that administrations of 10E8VLS alone and concurrently with VRC07-523LS will be well-tolerated in healthy adults. A secondary hypothesis was that both broadly neutralizing monoclonal antibodies (bNAbs) will be detectable in human sera with a definable half-life.

Product Description:

The 10E8VLS and VRC07-523LS bNAbs target the HIV-1 envelope at distinct epitopes: 10E8VLS recognizes the membrane proximal external region (MPER) and proximal viral membrane lipid of gp41, while VRC07-523LS recognizes the CD4 binding site of gp120. Both antibodies are human in origin, contain two amino acid modifications within the C-terminus of the heavy chain constant region designed to improve antibody half-life in vivo, and were developed by the VRC/NIAID/NIH. The 10E8VLS and VRC07-523LS bNAbs were manufactured under current Good Manufacturing Practice (cGMP) regulations at the VRC Pilot Plant operated under contract by the Vaccine Clinical Materials Program (VCMP), Leidos Biomedical Research, Inc., Frederick, MD.

The 10E8VLS drug product was supplied at a concentration of 100 mg/mL in a sterile, aqueous, buffered solution of 5.25 mL in single-use 10 mL glass vials. The VRC07-523LS drug product was supplied at a concentration of 100 mg/mL in an isotonic, sterile solution of 6.25 mL in single-use 10 mL glass vials. Each drug product was prepared for administration in separate syringes.

Participants:

Healthy adults, 18-60 years of age.

Study Plan:

This open-label study included 4 dosing regimens of either 10E8VLS (5 mg/kg) administered alone or 10E8VLS (5 mg/kg) and VRC07-523LS (5 mg/kg). All injections were administered by the subcutaneous (SC) route. For Groups 1 and 2, 10E8VLS was to be administered once or three-times at 12-week intervals. For Groups 3 and 4, 10E8VLS and VRC07-523LS were to be administered once or three-times at 12-week intervals, respectively. Enrollment began with Groups 1 and 2, followed by Groups 3 and 4.

VRC 610 Study Schema:

* Group 1; Study Product: 10E8VLS; Planned Participants per Group: 3; Dose Administered SC: 5 mg/kg; Day 0
* Group 2; Study Product: 10E8VLS; Planned Participants per Group: 3; Dose Administered SC: 5 mg/kg; Day 0, Week 12*, Week 24*
* Group 3 (a,b); Study Product: 10E8VLS+VRC07-523LS; Planned Participants per Group: 5; Dose Administered SC: 5 mg/kg of each MAb; Day 0
* Group 4 (a,b); Study Product: 10E8VLS+VRC07-523LS; Planned Participants per Group: 5; Dose Administered SC: 5 mg/kg of each MAb; Day 0, Week 12*, Week 24*
* Total Planned Participants = 16
* Total Actual Participants = 9 (c)

(*)Participants received only one product administration on Day 0 because of the voluntary study pause and termination by Investigational New Drug (IND) Sponsor/Principal Investigator (PI) decision.

1. Enrollment into Group 3 and 4 commenced after positive protocol safety review team (PSRT) review of safety data from Groups 1 and 2
2. 10E8VLS and VRC07-523LS were provided in separate syringes and administered at the same visit.
3. The expected enrollment was 16 participants; however, enrollment was voluntarily paused by the IND Sponsor/PI and the study ultimately stopped after several Grade 2 and Grade 3 redness local reactogenicity reactions were observed at 10E8VLS injection sites.

Study Duration:

Study participation was expected to be approximately 24 weeks for participants in Groups 1 and 3, and 48 weeks for participants in Groups 2 and 4. Participants in the repeat-dose groups (2 and 4) were converted to a modified schedule per protocol. Study participation for all participants was approximately 24 weeks after Day 0 product administration.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Willing and able to complete the informed consent process.
  2. 18 to 60 years of age.
  3. Based on history and examination, in good general health and without history of any of the conditions listed in the exclusion criteria.
  4. Willing to have blood samples collected, stored indefinitely, and used for research purposes.
  5. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
  6. Screening laboratory criteria within 84 days prior to enrollment must meet the following criteria:
* White blood cell count (WBC): 2,500-12,000/mm^3.
* WBC differential: Within institutional normal range or accompanied by the Principal Investigator (PI) or designee approval.
* Platelets: 125,000 - 400,000/mm^3.
* Hemoglobin: Within institutional normal range or accompanied by PI or designee approval.
* Creatinine: less than or equal to 1.1 x Upper Limit of Normal (ULN).
* Aspartate aminotransferase (AST): less than or equal to 1.25 x ULN
* Alanine aminotransferase (ALT): less than or equal to 1.25 x ULN.
* Negative for HIV infection by an FDA approved method of detection.
* Negative for Hepatitis B core antibody (HBcAb) and Hepatitis C virus antibody (HCV Ab).

Female-Specific Criteria:

7. If a woman is of reproductive potential and sexually active with a male partner, then she agrees to use an effective means of birth control from the time of study enrollment until the last study visit, or to be monogamous with a partner who has had a vasectomy.

8. Negative Beta-HCG (human chorionic gonadotropin) pregnancy test (urine or serum) on day of enrollment for women presumed to be of reproductive potential.

* EXCLUSION CRITERIA:

  1. Woman who is breast-feeding, or planning to become pregnant during the study.
  2. Prior receipt of licensed or investigational monoclonal antibody.
  3. Weight > 115 kg.
  4. Any history of a severe allergic reaction with generalized urticaria, angioedema or anaphylaxis within the 2 years prior to enrollment that has a reasonable risk of recurrence during the study.
  5. Hypertension that is not well controlled.
  6. Receipt of any investigational study agent within 28 days prior to enrollment.
  7. Any other chronic or clinically significant condition that in the opinion of investigator would jeopardize the safety or rights of the volunteer including (but not limited to): diabetes mellitus type I/II, chronic hepatitis; OR clinically significant forms of drug or alcohol abuse, asthma, autoimmune disease, psychiatric disorders, heart disease, or cancer.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2019-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin R Gaudinski, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang J, Ofek G, Laub L, Louder MK, Doria-Rose NA, Longo NS, Imamichi H, Bailer RT, Chakrabarti B, Sharma SK, Alam SM, Wang T, Yang Y, Zhang B, Migueles SA, Wyatt R, Haynes BF, Kwong PD, Mascola JR, Connors M. Broad and potent neutralization of HIV-1 by a gp41-specific human antibody. Nature. 2012 Nov 15;491(7424):406-12. doi: 10.1038/nature11544. Epub 2012 Sep 18. PMID 23151583
- [Background] Kwon YD, Georgiev IS, Ofek G, Zhang B, Asokan M, Bailer RT, Bao A, Caruso W, Chen X, Choe M, Druz A, Ko SY, Louder MK, McKee K, O'Dell S, Pegu A, Rudicell RS, Shi W, Wang K, Yang Y, Alger M, Bender MF, Carlton K, Cooper JW, Blinn J, Eudailey J, Lloyd K, Parks R, Alam SM, Haynes BF, Padte NN, Yu J, Ho DD, Huang J, Connors M, Schwartz RM, Mascola JR, Kwong PD. Optimization of the Solubility of HIV-1-Neutralizing Antibody 10E8 through Somatic Variation and Structure-Based Design. J Virol. 2016 Jun 10;90(13):5899-5914. doi: 10.1128/JVI.03246-15. Print 2016 Jul 1. PMID 27053554
- [Derived] Awan SF, Pegu A, Strom L, Carter CA, Hendel CS, Holman LA, Costner PJ, Trofymenko O, Dyer R, Gordon IJ, Rothwell RSS, Hickman SP, Conan-Cibotti M, Doria-Rose NA, Lin BC, O'Connell S, Narpala SR, Almasri CG, Liu C, Ko S, Kwon YD, Namboodiri AM, Pandey JP, Arnold FJ, Carlton K, Gall JG, Kwong PD, Capparelli EV, Bailer RT, McDermott AB, Chen GL, Koup RA, Mascola JR, Coates EE, Ledgerwood JE, Gaudinski MR; VRC 610 study team. Phase 1 trial evaluating safety and pharmacokinetics of HIV-1 broadly neutralizing mAbs 10E8VLS and VRC07-523LS. JCI Insight. 2024 Apr 8;9(7):e175375. doi: 10.1172/jci.insight.175375. PMID 38587079
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-I-0113.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 2: 10E8VLS (5 mg/kg) SC Multiple Dose Group* (*Only One Dose Received): 10E8VLS (5 mg/kg) administered by the SC route (Day 0, Week 12*, Week 24*)
  *Participants received only one product administration on Day 0 because of the voluntary study pause and termination by the IND Sponsor/PI decision.
  VRC-HIVMAB095-00-AB (10E8VLS): 10E8VLS is an investigational Monoclonal Antibody targeted to the membrane proximal external region and proximal viral membrane lipid region of HIV-1.
- Group 4: 10E8VLS+VRC07-523LS (5 mg/kg Each) SC Multiple Dose Group* (*Only One Dose Received): 10E8VLS (5 mg/kg)+VRC07-523LS (5 mg/kg) administered by the SC route (Day 0, Week 12*, Week 24*)
  *Participants received only one product administration on Day 0 because of the voluntary study pause and termination by the IND Sponsor/PI decision.
  VRC-HIVMAB095-00-AB (10E8VLS): 10E8VLS is an investigational Monoclonal Antibody targeted to the membrane proximal external region and proximal viral membrane lipid region of HIV-1.
  VRC-HIVMAB075-00-AB (VRC07-523LS): VRC07-523LS is an investigational Monoclonal Antibody targeted to the CD4 binding site of HIV-1.
Period: Overall Study
Arm/Group | Group 1: 10E8VLS (5 mg/kg) SC Single Dose Group | Group 2: 10E8VLS (5 mg/kg) SC Multiple Dose Group* (*Only One Dose Received) | Group 3: 10E8VLS+VRC07-523LS (5 mg/kg Each) SC Single Dose Group | Group 4: 10E8VLS+VRC07-523LS (5 mg/kg Each) SC Multiple Dose Group* (*Only One Dose Received)
Started | 3 | 3 | 1 | 2
Product Administration Completed | 3 | 0 | 1 | 0
Discontinued Product Administrations (All altered or discontinued product administration schedules were due to the IND Sponsor/PI decision to terminate the study.) | 0 | 3 | 0 | 2 (One Group 4 participant enrolled but did not receive product due to IND/PI voluntary study pause.)
Completed | 3 | 3 | 1 | 1
Not Completed | 0 | 0 | 0 | 1
Not completed — IND Sponsor/PI Voluntary Study Pause | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Population includes all enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: 10E8VLS (5 mg/kg) SC Single Dose Group | Group 2: 10E8VLS (5 mg/kg) SC Multiple Dose Group* (*Only One Dose Received) | Group 3: 10E8VLS+VRC07-523LS (5 mg/kg Each) SC Single Dose Group | Group 4: 10E8VLS+VRC07-523LS (5 mg/kg Each) SC Multiple Dose Group* (*Only One Dose Received) | Total
Number analyzed (Participants) | 3 | 3 | 1 | 2 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.7 (16.1) | 27.7 (5.0) | 40.0 (0.0) | 45.0 (15.6) | 33.6 (12.6)
Age, Customized [Count of Participants; unit: Participants]
  18-20 years | 1 | 0 | 0 | 0 | 1
  21-30 years | 1 | 2 | 0 | 0 | 3
  31-40 years | 0 | 1 | 1 | 1 | 3
  41-50 years | 1 | 0 | 0 | 0 | 1
  51-60 years | 0 | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 0 | 1 | 3
  Male | 1 | 3 | 1 | 1 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 0 | 0 | 1
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 1 | 3 | 1 | 2 | 7
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
Weight (kg) [Mean (Standard Deviation); unit: kilograms] | 81.7 (15.1) | 80.1 (18.4) | 91.1 (0.0) | 75.7 (1.3) | 80.9 (12.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms Within 3 Days of Product Administration
Description: Local symptoms were recorded by participants using a 3-day diary. Solicited local symptoms include pain/tenderness, bruising, redness, swelling, and pruritus (itchiness) at the product administration site. Clinicians reviewed the diary with the participant and collected resolution information for any symptoms that were not resolved within 3 days. Participants were counted once for each symptom at the worst severity if they experienced the symptom at any severity during the reporting period. The number reported for "Any Local Symptom" is the number of participants reporting any local symptom at the worst severity. Reactogenicity grading was done by Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1.
Time Frame: 3 days after product administration
Population: Participants in Groups 1 and 2 (N=6) received 10E8VLS and Groups 3 and 4 (N=2) received 10E8VLS+VRC07-523LS. Participants in Groups 2 and 4 were assigned to receive 3 repeat product administrations but received only 1 due to the voluntary termination of study product administration by the IND sponsor. The 2nd and 3rd doses for the 3 Group 2 participants assigned to receive 10E8VLS, and the single Group 4 participant assigned to receive 10E8VLS+VRC07-523LS were not administered.
Measure: Count of Participants; unit: Participants
Groups:
- Overall 10E8VLS Groups: Total number of participants who received an SC injection of 10E8VLS alone - Groups 1 and 2 only received 10E8VLS
- Group 3: 10E8VLS Site Only in 10E8VLS+VRC07-523LS (5 mg/kg) SC Single Dose Group; Group 3: VRC07-523LS Site Only in 10E8VLS+VRC07-523LS (5 mg/kg) SC Single Dose Group: 10E8VLS (5 mg/kg)+VRC07-523LS (5 mg/kg) administered by the SC route (Day 0)
  VRC-HIVMAB095-00-AB (10E8VLS): 10E8VLS is an investigational Monoclonal Antibody targeted to the membrane proximal external region and proximal viral membrane lipid region of HIV-1.
  VRC-HIVMAB075-00-AB (VRC07-523LS): VRC07-523LS is an investigational Monoclonal Antibody targeted to the CD4 binding site of HIV-1.
- Group 4: 10E8VLS Site Only in 10E8VLS+VRC07-523LS (5 mg/kg) SC Multiple Dose Group* (*Only 1 Dose); Group 4: VRC07-523LS Site Only- 10E8VLS+VRC07-523LS (5 mg/kg) SC Multiple Dose Group* (*Only 1 Dose): 10E8VLS (5 mg/kg)+VRC07-523LS (5 mg/kg) administered by the SC route (Day 0, Week 12*, Week 24*)
  *Participants received only one product administration on Day 0 because of the voluntary study pause and termination by the IND Sponsor/PI decision.
  VRC-HIVMAB095-00-AB (10E8VLS): 10E8VLS is an investigational Monoclonal Antibody targeted to the membrane proximal external region and proximal viral membrane lipid region of HIV-1.
  VRC-HIVMAB075-00-AB (VRC07-523LS): VRC07-523LS is an investigational Monoclonal Antibody targeted to the CD4 binding site of HIV-1.
- Overall 10E8VLS Site Only in 10E8VLS+VRC07-523LS Groups: Total number of participants who received an SC injection of 10E8VLS in Groups 3 and 4 who received 10E8VLS and VRC07-523LS concurrently
- Overall VRC07-523LS Site Only in 10E8VLS+VRC07-523LS Groups: Total number of participants who received an SC injection of VRC07-523LS in Groups 3 and 4 who received 10E8VLS and VRC07-523LS concurrently
Arm/Group | Group 1: 10E8VLS (5 mg/kg) SC Single Dose Group | Group 2: 10E8VLS (5 mg/kg) SC Multiple Dose Group* (*Only One Dose Received) | Overall 10E8VLS Groups | Group 3: 10E8VLS Site Only in 10E8VLS+VRC07-523LS (5 mg/kg) SC Single Dose Group | Group 4: 10E8VLS Site Only in 10E8VLS+VRC07-523LS (5 mg/kg) SC Multiple Dose Group* (*Only 1 Dose) | Overall 10E8VLS Site Only in 10E8VLS+VRC07-523LS Groups | Group 3: VRC07-523LS Site Only in 10E8VLS+VRC07-523LS (5 mg/kg) SC Single Dose Group | Group 4: VRC07-523LS Site Only- 10E8VLS+VRC07-523LS (5 mg/kg) SC Multiple Dose Group* (*Only 1 Dose) | Overall VRC07-523LS Site Only in 10E8VLS+VRC07-523LS Groups
Number analyzed (Participants) | 3 | 3 | 6 | 1 | 1 | 2 | 1 | 1 | 2
Participants
  Pain/Tenderness: None | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Pain/Tenderness: Mild | 3 | 3 | 6 | 1 | 1 | 2 | 0 | 0 | 0
  Pain/Tenderness: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Tenderness: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bruising: None | 2 | 2 | 4 | 1 | 1 | 2 | 1 | 1 | 2
  Bruising: Mild | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Bruising: Moderate | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Bruising: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Redness: None | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Redness: Mild | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
  Redness: Moderate | 2 | 2 | 4 | 0 | 1 | 1 | 1 | 0 | 1
  Redness: Severe | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Swelling: None | 0 | 3 | 3 | 0 | 0 | 0 | 1 | 1 | 2
  Swelling: Mild | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
  Swelling: Moderate | 2 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0
  Swelling: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pruritus: None | 3 | 2 | 5 | 1 | 1 | 2 | 1 | 1 | 2
  Pruritus: Mild | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Pruritus: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pruritus: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Local Symptom Reported: None | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Local Symptom Reported: Mild | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 1
  Any Local Symptom Reported: Moderate | 2 | 2 | 4 | 0 | 1 | 1 | 1 | 0 | 1
  Any Local Symptom Reported: Severe | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms Within 3 Days of Product Administration
Description: Participants recorded 3-day systemic symptoms in a diary after each study product administration. Solicited systemic symptoms include: unusually tired/feeling unwell, muscles aches, headache, chills, nausea, temperature and joint pain. Participants recorded highest measured temperature daily. Clinicians reviewed the diary with the participant and collected resolution information for any symptoms that were not resolved within 3 days. Participants were counted once for each symptom at the worst severity if they indicated experiencing the symptom at any severity during the reporting period. The number reported for "Any Systemic Symptom" is the number of participants reporting any systemic symptom at the worst severity. Reactogenicity grading was done by Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1.
Time Frame: 3 days after product administration
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Group 4: 10E8VLS+VRC07-523LS (5 mg/kg Each) SC Multiple Dose Group* (*Only 1 Dose): 10E8VLS (5 mg/kg)+VRC07-523LS (5 mg/kg) administered by the SC route (Day 0, Week 12*, Week 24*)
  *Participants received only one product administration on Day 0 because of the voluntary study pause and termination by the IND Sponsor/PI decision.
  VRC-HIVMAB095-00-AB (10E8VLS): 10E8VLS is an investigational Monoclonal Antibody targeted to the membrane proximal external region and proximal viral membrane lipid region of HIV-1.
  VRC-HIVMAB075-00-AB (VRC07-523LS): VRC07-523LS is an investigational Monoclonal Antibody targeted to the CD4 binding site of HIV-1.
- Overall 10E8VLS+VRC07-523LS Groups: Total number of participants who received an SC injection of 10E8VLS and an SC injection of VRC07-523LS concurrently - Groups 3 and 4 received 10E8VLS and VRC07-523LS
Arm/Group | Group 1: 10E8VLS (5 mg/kg) SC Single Dose Group | Group 2: 10E8VLS (5 mg/kg) SC Multiple Dose Group* (*Only One Dose Received) | Overall 10E8VLS Groups | Group 3: 10E8VLS+VRC07-523LS (5 mg/kg Each) SC Single Dose Group | Group 4: 10E8VLS+VRC07-523LS (5 mg/kg Each) SC Multiple Dose Group* (*Only 1 Dose) | Overall 10E8VLS+VRC07-523LS Groups
Number analyzed (Participants) | 3 | 3 | 6 | 1 | 1 | 2
Participants
  Malaise: None | 2 | 3 | 5 | 0 | 1 | 1
  Malaise: Mild | 1 | 0 | 1 | 1 | 0 | 1
  Malaise: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Malaise: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: None | 3 | 2 | 5 | 0 | 1 | 1
  Myalgia: Mild | 0 | 1 | 1 | 1 | 0 | 1
  Myalgia: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Headache: None | 3 | 3 | 6 | 1 | 1 | 2
  Headache: Mild | 0 | 0 | 0 | 0 | 0 | 0
  Headache: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Headache: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Chills: None | 3 | 3 | 6 | 0 | 1 | 1
  Chills: Mild | 0 | 0 | 0 | 1 | 0 | 1
  Chills: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Chills: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: None | 2 | 3 | 5 | 0 | 1 | 1
  Nausea: Mild | 1 | 0 | 1 | 1 | 0 | 1
  Nausea: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: None | 3 | 3 | 6 | 0 | 1 | 1
  Temperature: Mild | 0 | 0 | 0 | 1 | 0 | 1
  Temperature: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Joint Pain: None | 3 | 3 | 6 | 0 | 1 | 1
  Joint Pain: Mild | 0 | 0 | 0 | 1 | 0 | 1
  Joint Pain: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Joint Pain: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Any Systemic Symptom: None | 2 | 2 | 4 | 0 | 1 | 1
  Any Systemic Symptom: Mild | 1 | 1 | 2 | 1 | 0 | 1
  Any Systemic Symptom: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Any Systemic Symptom: Severe | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With One or More Unsolicited Non-Serious Adverse Events
Description: Unsolicited adverse events (AEs) collected during the period from study product administration at Day 0 through 56 days after product administration. After the indicated time period through the last expected study visit at 24 weeks after product administration, only new chronic medical conditions collected as unsolicited AEs. The number reported is the number of participants who experienced at least one AE in the reporting period. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Up to 24 weeks after product administration
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Group 4: 10E8VLS+VRC07-523LS (5 mg/kg Each) SC Multiple Dose Group* (*Only One Dose Received): 10E8VLS (5 mg/kg)+VRC07-523LS (5 mg/kg each) administered by the SC route (Day 0, Week 12*, Week 24*)
  *Participants received only one product administration on Day 0 because of the voluntary study pause and termination by the IND Sponsor/PI decision.
  VRC-HIVMAB095-00-AB (10E8VLS): 10E8VLS is an investigational Monoclonal Antibody targeted to the membrane proximal external region and proximal viral membrane lipid region of HIV-1.
  VRC-HIVMAB075-00-AB (VRC07-523LS): VRC07-523LS is an investigational Monoclonal Antibody targeted to the CD4 binding site of HIV-1.
- Overall: Total number of participants who received 10E8VLS administered alone or concurrently with VRC07-523LS
Arm/Group | Group 1: 10E8VLS (5 mg/kg) SC Single Dose Group | Group 2: 10E8VLS (5 mg/kg) SC Multiple Dose Group* (*Only One Dose Received) | Group 3: 10E8VLS+VRC07-523LS (5 mg/kg Each) SC Single Dose Group | Group 4: 10E8VLS+VRC07-523LS (5 mg/kg Each) SC Multiple Dose Group* (*Only One Dose Received) | Overall
Number analyzed (Participants) | 3 | 3 | 1 | 1 | 8
Participants
  Related to 10E8VLS | 0 | 0 | 0 | 0 | 0
  Related to VRC07-523LS | 0 | 0 | 1 | 0 | 1
  Unrelated to 10E8VLS or VRC07-523LS | 2 | 2 | 0 | 0 | 4

4. Primary Outcome: Number of Participants With Serious Adverse Events
Description: Serious adverse events (SAEs) collected during the period from study product administration at Day 0 through 24 weeks after the product administration.
Time Frame: Up to 24 weeks after product administration
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 10E8VLS (5 mg/kg) SC Single Dose Group | Group 2: 10E8VLS (5 mg/kg) SC Multiple Dose Group* (*Only One Dose Received) | Group 3: 10E8VLS+VRC07-523LS (5 mg/kg Each) SC Single Dose Group | Group 4: 10E8VLS+VRC07-523LS (5 mg/kg Each) SC Multiple Dose Group* (*Only One Dose Received) | Overall
Number analyzed (Participants) | 3 | 3 | 1 | 1 | 8
Participants | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of 10E8VLS Administered Alone or Concurrently With VRC07-523LS
Description: Cmax is the peak serum concentration that 10E8VLS achieves after it has been administered: it is determined as maximum value on the summary pharmacokinetic (PK) curve for the overall study population.
  Serum was collected at the following time points: Groups 1 and 3: Pre-injection (baseline), and 24, 48 and 72 hours post injection, followed by Weeks 1-4, 8, 12, 16, 20 and 24 post-injection; Groups 2 and 4: Pre-injection (baseline), and 24, 48 and 72 hours post injection, and Weeks 1, 2, 4, 8, 12-14, 16, 20 and 24 post injection
Time Frame: Up to 24 weeks after product administration
Population: Participants received 10E8VLS administered alone or concurrently with VRC07-523LS (N=8), where "N" signifies the number analyzed. The overall population (N=8) was analyzed for this measure as all study groups received only one 10E8VLS administration. Due to voluntary termination of study product administration by the IND sponsor, 2nd and 3rd administrations for the 3 participants assigned to receive 10E8VLS, and the one participant assigned to receive 10E8VLS+VRC07-523LS were not administered.
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- All 10E8VLS 5 mg/kg SC Groups (With or Without VRC07-523LS): Total number of participants who received 10E8VLS administered alone or concurrently with VRC07-523LS
Arm/Group | All 10E8VLS 5 mg/kg SC Groups (With or Without VRC07-523LS)
Number analyzed (Participants) | 8
µg/mL | 28.3 (11.1)

6. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax) of 10E8VLS Administered Alone or Concurrently With VRC07-523LS
Description: Tmax is the time it takes to reach Cmax of 10E8VLS after it has been administered; it is determined based on the summary PK curve for the overall study population.
  Serum was collected at the following time points: Groups 1 and 3: Pre-injection (baseline), and 24, 48 and 72 hours post injection, followed by Weeks 1-4, 8, 12, 16, 20 and 24 post-injection; Groups 2 and 4: Pre-injection (baseline), and 24, 48 and 72 hours post injection, and Weeks 1, 2, 4, 8, 12-14, 16, 20 and 24 post injection
Time Frame: Up to 24 weeks after product administration
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: days
Arm/Group | All 10E8VLS 5 mg/kg SC Groups (With or Without VRC07-523LS)
Number analyzed (Participants) | 8
days | 2.6 (0.5)

7. Secondary Outcome: Area Under the Curve (AUC0-28D) of 10E8VLS Administered Alone or Concurrently With VRC07-523LS
Description: The AUC0-28D represents the total drug exposure in 28 days after 10E8VLS administration; it is determined based on the summary PK curve for the overall study population.
  Serum was collected at the following time points: Groups 1 and 3: Pre-injection (baseline), and 24, 48 and 72 hours post injection, followed by Weeks 1, 2, 3 and 4 post injection; Groups 2 and 4: Pre-injection (baseline) and 24, 48 and 72 hours post injection and Weeks 1, 2 and 4 post injection.
Time Frame: Administration (0h) up to 28 days after product administration
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: µg*d/mL
Arm/Group | All 10E8VLS 5 mg/kg SC Groups (With or Without VRC07-523LS)
Number analyzed (Participants) | 8
µg*d/mL | 322 (114)

8. Secondary Outcome: 4 Week Mean Serum Concentration of 10E8VLS Administered Alone or Concurrently With VRC07-523LS
Description: The mean of individual participant 10E8VLS serum concentrations. The overall population was analyzed as all participants received only one 10E8VLS administration.
Time Frame: Administration (0h) up to 28 days after product administration
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | All 10E8VLS 5 mg/kg SC Groups (With or Without VRC07-523LS)
Number analyzed (Participants) | 8
µg/mL | 3.06 (1.22)

9. Secondary Outcome: Clearance Rate of 10E8VLS Administered Alone or Concurrently With VRC07-523LS
Description: Rate of 10E8VLS elimination divided by the plasma 10E8VLS concentration; determined based on the summary PK curve for the overall study population.
  Serum was collected at the following time points: Groups 1 and 3: Pre-injection (baseline), and 24, 48 and 72 hours post injection, followed by Weeks 1, 2, 3 and 4 post injection; Groups 2 and 4: Pre-injection (baseline) and 24, 48 and 72 hours post injection and Weeks 1, 2 and 4 post injection.
Time Frame: Administration (0h) up to 28 days after product administration
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mL/d
Arm/Group | All 10E8VLS 5 mg/kg SC Groups (With or Without VRC07-523LS)
Number analyzed (Participants) | 8
mL/d | 1309 (496)

10. Secondary Outcome: Overall Half-Life (T1/2) of 10E8VLS Administered Alone or Concurrently With VRC07-523LS
Description: Half-life (T1/2) is the time required for half of the drug to be eliminated from the serum.
  Serum was collected at the following time points: Groups 1 and 3: Pre-injection (baseline), and 24, 48 and 72 hours post injection, followed by Weeks 1, 2, 3 and 4 post injection; Groups 2 and 4: Pre-injection (baseline) and 24, 48 and 72 hours post injection and Weeks 1, 2 and 4 post injection.
Time Frame: Administration (0h) up to 28 days after product administration
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: days
Arm/Group | All 10E8VLS 5 mg/kg SC Groups (With or Without VRC07-523LS)
Number analyzed (Participants) | 8
days | 8.1 (1.5)

ADVERSE EVENTS:
Time Frame: Solicited adverse events (AEs) included local administration site and systemic AEs reported by participants at the worst severity through 3 days after the product administration. Unsolicited AEs were reported from the date of product administration through 56 days thereafter, and new chronic medical conditions and SAEs with onset any time following the date of last product administration through 24 weeks.
Description: Solicited AEs collected through systematic assessment and unsolicited AEs collected through non-systematic assessment represent the number and percentage of participants reporting the event. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Arm/Group | Group 1: 10E8VLS (5 mg/kg) SC Single Dose Group | Group 2: 10E8VLS (5 mg/kg) SC Multiple Dose Group* (*Only One Dose Received) | Group 3: 10E8VLS+VRC07-523LS (5 mg/kg Each) SC Single Dose Group | Group 4: 10E8VLS+VRC07-523LS (5 mg/kg Each) SC Multiple Dose Group* (*Only One Dose Received)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 1/1 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: 10E8VLS (5 mg/kg) SC Single Dose Group (N=3) | Group 2: 10E8VLS (5 mg/kg) SC Multiple Dose Group* (*Only One Dose Received) (N=3) | Group 3: 10E8VLS+VRC07-523LS (5 mg/kg Each) SC Single Dose Group (N=1) | Group 4: 10E8VLS+VRC07-523LS (5 mg/kg Each) SC Multiple Dose Group* (*Only One Dose Received) (N=1)
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Administration site [10E8VLS] bruising (General disorders) | 1 | 1 | 0 | 0
Administration site [10E8VLS] erythema (General disorders) | 2 | 3 | 1 | 1 — Redness
Administration site [10E8VLS] pain/tenderness (General disorders) | 3 | 3 | 1 | 1
Administration site [10E8VLS] pruritis (General disorders) | 0 | 1 | 0 | 0 — Itching
Administration site [10E8VLS] swelling (General disorders) | 3 | 0 | 1 | 1
Administration site [VRC07-523LS] erythema (General disorders) | 0 | 0 | 1 | 1 — Redness
Chills (General disorders) | 0 | 0 | 1 | 0
Injection site [VRC07-523LS site] erythema (General disorders) | 0 | 0 | 1 | 0 — Redness
Malaise (General disorders) | 1 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 — Temperature (Fever)
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 — Joint pain
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study never resumed after the voluntary pause. Participants in the repeat-dose groups (2 and 4) were converted to a modified schedule per protocol. Study participation for all participants was approximately 24 weeks after Day 0 product administration. The overall population (N=8) was analyzed for the pharmacokinetic (PK) outcome measures as all study groups received only one 10E8VLS administration. Small group size has not allowed for meaningful PK analysis of each group separately.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-09-12): https://cdn.clinicaltrials.gov/large-docs/15/NCT03565315/Prot_SAP_ICF_000.pdf